CLINICAL TRIAL: NCT03849768
Title: A Phase III Randomized, Controlled, Double-Blind, Multicenter Clinical Trial to Evaluate the Efficacy and Safety of HS-10296 Versus Gefitinib as First-Line Therapy for Locally Advanced or Metastatic NSCLC With EGFR Sensitizing Mutations
Brief Title: A Study to Evaluate Safety and Efficacy of HS-10296 as First-Line Treatment in Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-10296-03-01
Record Dates: First submitted 2018-11-23; First posted 2019-02-21 (Actual); Results first posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2022-10

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aumolertinib; Gefitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HS-10296 (Experimental): 110mg PO once daily
  Interventions: Drug: HS-10296
- Gefitinib (Active Comparator): 250mg PO once daily
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: HS-10296 — Drug: HS-10296 110 mg/55 mg + placebo The initial dose of HS-10296 110 mg once daily can be reduced to 55 mg once daily under specific circumstances. A cycle of treatment is defined as 21 days of once daily treatment. Number of Cycles: as long as patients are continuing to show clinical benefit, as judged by the Investigator, and in the absence of discontinuation criteria.
  Other Names: Investigational Product
  Arms: HS-10296
Drug: Gefitinib — Drug: Gefitinib 250 mg + placebo The initial dose of Gefitinib 250 mg once daily cannot be reduced. A cycle of treatment is defined as 21 days of once daily treatment. Number of cycles: as long as patients are continuing to show clinical benefit, as judged by the Investigator, and in the absence of discontinuation criteria.
  Other Names: Comparator Product
  Arms: Gefitinib

SUMMARY:
This is a randomized, controlled, double-blind, multicenter, phase III clinical study.

DETAILED DESCRIPTION:
This is a randomized, controlled, double-blind, multicenter, phase III clinical trial, evaluating the efficacy and safety of HS-10296 compared to gefitinib in patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) with epidermal growth factor receptor sensitizing mutations (EGFRm+) who have not received systemic therapy. Patients are randomly assigned to an HS-10296 treatment group or a gefitinib treatment group at a ratio of 1:1 and receive a once-daily oral dose of HS-10296 or gefitinib, in order to compare the efficacy and safety of the two different treatment regimens.

ELIGIBILITY:
Inclusion Criteria: Inclusion Criteria:

Any patient who meets all of the following inclusion criteria will qualify for entry into the study:

1. Provision of informed consent prior to any study specific procedures, sampling and analyses.
2. Male or female, age at least 18 years.
3. Pathologically confirmed locally advanced or metastatic NSCLC (e.g. this may occur systemic recurrence after prior surgery for early stage disease or patients may be newly diagnosed with stage IIIB/IV disease). Patients must be treatment-naïve for locally advanced or metastatic NSCLC. Prior adjuvant and neo-adjuvant therapy is permitted (chemotherapy, radiotherapy, investigational agents) provided all other entry criteria are satisfied.
4. The tumour harbours one of the 2 common EGFR mutations known to be associated with EGFR-TKI sensitivity (Ex19del, L858R), either or in combination with other EGFR mutations assessed by central testing using tumour tissue sample or blood sample.
5. A WHO performance status equal to 0-1 with no deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks.
6. At least 1 lesion that has not previously been irradiated, that has not been chosen for biopsy during the study screening period, and that can be accurately measured at Baseline as ≥ 10 mm in the longest diameter (except lymph nodes, which must have short axis ≥ 15mm) with computerized tomography (CT) or magnetic resonance imaging (MRI), whichever is suitable for accurately repeated measurements. If only one measurable lesion exists, it is acceptable to be used (as a target lesion) as long as it has not been previously irradiated and baseline tumour assessment scans are done at least 14days afar the screening biopsy is performed.
7. Females should be using adequate contraceptive measures throughout the study; should not be breastfeeding at the time of screening, during the study and until 3 months after completion of the study; and must have a negative pregnancy test prior to start of dosing if of childbearing potential or must have evidence of non-childbearing potential by fulfilling 1 of the following criteria at Screening:

   1. Postmenopausal defined as age more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments.
   2. Women under 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more, following cessation of exogenous hormonal treatments, and with luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the postmenopausal range for the laboratory.
   3. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, but not by tubal ligation.
8. Male patients should be willing to use barrier contraception (i.e., condoms).
9. For inclusion in study, patient must provide a written informed consent.

   -

Exclusion Criteria: Exclusion Criteria:

Any patient who meets any of the following exclusion criteria will not qualify for entry into the study:

1. Treatment with any of the following:

   1. Prior treatment with systemic anti-cancer therapy for locally advancer or metastatic NSCLC including chemotherapy, biologic therapy, immunotherapy, or any investigational drug.
   2. Prior treatment with an EGFR TKI.
   3. Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study drug.
   4. Radiotherapy with a limited field of radiation for palliation within 4 week of the first dose of study drug, with the exception of patients receiving radiation to > 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug.
   5. Medications that are predominantly CYP3A4 strong inhibitors or inducers or sensitive substrates of CYP3A4 with a narrow therapeutic range within 7 days of the first dose of study drug.
2. Any concurrent and/or other active malignancy that has required treatment within 2 years of first dose of study drug.
3. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 at the time of starting study treatment, with the exception of alopecia and Grade 2, prior platinum-therapy related neuropathy.
4. Spinal cord compression or brain metastases unless asymptomatic, stable, and not requiring steroids for at least 2 weeks prior to start of study treatment.
5. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension or active bleeding diatheses, which, in the Investigator's opinion, makes it undesirable for the patient to participate in the trial OR which would jeopardize compliance with the protocol such as active infection. Screening for chronic conditions is not required.
6. Refractory nausea, vomiting, or chronic gastrointestinal diseases, inability to swallow the study drug, or previous significant bowel resection that would preclude adequate absorption of HS 10296.
7. Any of the following cardiac criteria:

   1. Mean resting corrected QT interval (QTc) > 470 ms obtained from 3 electrocardiograms (ECGs), using the screening clinic's ECG machine and Fridericia's formula for QT interval correction (QTcF).
   2. Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG (e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval > 250 ms).
   3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval.
   4. Left ventricular ejection fraction (LVEF) ≤ 40%.
8. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis that required steroid treatment, or any evidence of clinically active interstitial lung disease.
9. Inadequate bone marrow reserve or organ function, as demonstrated by any of the following laboratory values:

   1. Absolute neutrophil count (ANC) <1.5×109 / L
   2. Platelet count <100×109 / L
   3. Hemoglobin <90 g/L（<9 g/dL）
   4. Alanine aminotransferase > 2.5 × upper limit of normal (ULN) if no demonstrable liver metastases or > 5 × ULN in the presence of liver metastases.
   5. Aspartate aminotransferase (AST) > 2.5 × ULN if no demonstrable liver metastases or > 5 × ULN in the presence of liver metastases.
   6. Total bilirubin (TBL) > 1.5 × ULN if no liver metastases or > 3 × ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases.
   7. Creatinine > 1.5 × ULN concurrent with creatinine clearance < 50 mL/min (measured or calculated by the Cockcroft-Gault equation); confirmation of creatinine clearance is only required when creatinine is > 1.5 × ULN.
10. Women who are breastfeeding or have a positive urine or serum pregnancy test at the Screening Visit.
11. History of hypersensitivity to any active or inactive ingredient of HS 10296 or to drugs with a similar chemical structure or class to HS 10296.
12. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
13. Any severe and uncontrolled ocular disease that may, in the ophthalmologist's opinion, present a specific risk to the patient's safety.
14. Any disease or condition that, in the opinion of the Investigator, would compromise the safety of the patient or interfere with study assessments.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 429 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2023-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Maniam Ajit, MD, Study Chair — Pacific Cancer Medical Center, Inc.
Locations (1):
- Beijing Cancer Hospital, Beijing, China

REFERENCES:
- [Derived] Lu S, Dong X, Jian H, Chen J, Chen G, Sun Y, Ji Y, Wang Z, Shi J, Lu J, Chen S, Lv D, Zhang G, Liu C, Li J, Yu X, Lin Z, Yu Z, Wang Z, Cui J, Xu X, Fang J, Feng J, Xu Z, Ma R, Hu J, Yang N, Zhou X, Wu X, Hu C, Zhang Z, Lu Y, Hu Y, Jiang L, Wang Q, Guo R, Zhou J, Li B, Hu C, Tong W, Zhang H, Ma L, Chen Y, Jie Z, Yao Y, Zhang L, Weng J, Li W, Xiong J, Ye X, Duan J, Yang H, Sun M, Wei H, Wei J, Zhang Z, Wu Q. Central nervous system efficacy of aumolertinib versus gefitinib in patients with untreated, EGFR-mutated, advanced non-small cell lung cancer: data from a randomized phase III trial (AENEAS). Cancer Commun (Lond). 2024 Sep;44(9):1005-1017. doi: 10.1002/cac2.12594. Epub 2024 Jul 17. PMID 39016053
- [Derived] Lu S, Dong X, Jian H, Chen J, Chen G, Sun Y, Ji Y, Wang Z, Shi J, Lu J, Chen S, Lv D, Zhang G, Liu C, Li J, Yu X, Lin Z, Yu Z, Wang Z, Cui J, Xu X, Fang J, Feng J, Xu Z, Ma R, Hu J, Yang N, Zhou X, Wu X, Hu C, Zhang Z, Lu Y, Hu Y, Jiang L, Wang Q, Guo R, Zhou J, Li B, Hu C, Tong W, Zhang H, Ma L, Chen Y, Jie Z, Yao Y, Zhang L, Jie W, Li W, Xiong J, Ye X, Duan J, Yang H, Sun M, Sun C, Wei H, Li C, Ali SM, Miller VA, Wu Q. AENEAS: A Randomized Phase III Trial of Aumolertinib Versus Gefitinib as First-Line Therapy for Locally Advanced or MetastaticNon-Small-Cell Lung Cancer With EGFR Exon 19 Deletion or L858R Mutations. J Clin Oncol. 2022 Sep 20;40(27):3162-3171. doi: 10.1200/JCO.21.02641. Epub 2022 May 17. PMID 35580297

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 429 participants were randomized to at 53 study sites.
Period: Overall Study
Arm/Group | HS-10296 | Gefitinib
Started | 214 | 215
Completed | 121 | 181
Not Completed | 93 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HS-10296 | Gefitinib | Total
Number analyzed (Participants) | 214 | 215 | 429
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 155 | 139 | 294
  >=65 years | 59 | 76 | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (9.59) | 60.6 (9.72) | 59.3 (9.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 135 | 269
  Male | 80 | 80 | 160
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 214 | 215 | 429
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Smoking status [Count of Participants; unit: Participants]
  Never smoked | 156 | 144 | 300
  smoked | 58 | 71 | 129

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of first dose until the date of radiological disease progression or until death due to any cause, based on the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, as assessed by investigators. Progression is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From baseline, then every 6 weeks, until disease progression or discontinuation from study. From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, approximately 2 years.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | HS-10296 | Gefitinib
Number analyzed (Participants) | 214 | 215
months | 19.3 [17.8 to 20.8] | 9.9 [8.3 to 12.6]

2. Secondary Outcome: Percentage of Participants With Objective Response Rate (ORR)
Description: ORR is defined as the percentage of patients who have at least 1 response of CR or PR prior to any evidence of progression. Target lesions and assessed by CT per RECIST v1.1 (Complete Response(CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.).
Time Frame: From baseline, then every 6 weeks, until disease progression or discontinuation from study.（up to 24 months）
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HS-10296 | Gefitinib
Number analyzed (Participants) | 214 | 215
percentage of participants | 73.8 [67.4 to 79.6] | 72.1 [65.6 to 78.0]

3. Secondary Outcome: Assess the Anti-tumor Activity: Duration of Response (DoR)
Description: DoR is defined as the time from the date of first documented response until the date of documented progression or death in the absence of disease progression assessed up to 24 months.
Time Frame: From baseline, then every 6 weeks, until disease progression or discontinuation from study. (up to 24 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | HS-10296 | Gefitinib
Number analyzed (Participants) | 214 | 215
months | 18.1 [15.2 to NA] — This outcome measure data was not available at the analysis cut-off due to insufficient number of participants with events. | 8.3 [6.9 to 11.1]

4. Secondary Outcome: Assess the Anti-tumor Activity: Disease Control Rate (DCR)
Description: The DCR is defined as the proportion of patients with a best overall response of CR, PR, or SD assessed up to 24 months.
Time Frame: From baseline, then every 6 weeks, until disease progression or discontinuation from study.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | HS-10296 | Gefitinib
Number analyzed (Participants) | 214 | 215
percentage | 93.0 [88.7 to 96.0] | 96.7 [93.4 to 98.7]

5. Secondary Outcome: Assess the Anti-tumor Activity: Depth of Response (DepOR)
Description: DepOR is defined as the percentage change in tumor shrinkage, based on longest diameter or reconstructed volume, observed at the lowest point (nadir) compared with baseline.
Time Frame: From baseline, then every 6 weeks, until disease progression or discontinuation from study.（up to 24 months）
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | HS-10296 | Gefitinib
Number analyzed (Participants) | 214 | 215
percentage of change from baseline | -44.95 (21.961) | -41.95 (19.966)

6. Secondary Outcome: Number of Participants With Adverse Events (AEs)/Serious Adverse Events (SAEs)
Description: Safety was assessed by AEs, which included abnormalities identified during a medical test (e.g. laboratory tests, vital signs, electrocardiogram, etc.) if the abnormality induced clinical signs or symptoms, needed active intervention, interruption or discontinuation of study medication or was clinically significant. A treatment-emergent AE (TEAE) was defined as an AE observed after starting administration of the study drug. AEs were considered serious (SAEs) if the AE resulted in death, was life threatening, resulted in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, resulted in congenital anomaly, or birth defect or required inpatient hospitalization or led to prolongation of hospitalization.
Time Frame: Continuously throughout the study until 28 days after HS-10296 discontinuation.From first dose of study drug up to 28 days after last dose of study drug taken (up to data cut-off (15 Jan 2021)),approximately 2 years.
Measure: Count of Participants; unit: Participants
Arm/Group | HS-10296 | Gefitinib
Number analyzed (Participants) | 214 | 215
Participants | 211 | 213

7. Secondary Outcome: Number of Participants With Dose Interruptions
Description: Participants had at least one delay in planned treatment due to treatment emergent adverse events.
Time Frame: From baseline, then every 6 weeks, until disease progression or discontinuation from study. (up to 24 months)
Measure: Count of Participants; unit: Participants
Arm/Group | HS-10296 | Gefitinib
Number analyzed (Participants) | 214 | 215
Participants | 36 | 53

8. Secondary Outcome: Number of Participants With Dose Reductions
Description: Participants had at least one reduction in planned treatment dosage due to treatment emergent adverse events. Every participant took 2 pills of HS
  -10296 + 1 pill of placebo(experimental arm) or 2pills of placebo + 1pill of Gefitinib (control arm). When a dose reduction was decided by INV, the set of "2 pills of placebo" was decreased resulting in no reduction of active compound in control arm, compliance with dose modification for AEs in Gefitinib's label which includes interruption, discontinuation but reduction.
Time Frame: From baseline, then every 6 weeks, until disease progression or discontinuation from study. (up to 24 months)
Measure: Count of Participants; unit: Participants
Arm/Group | HS-10296 | Gefitinib
Number analyzed (Participants) | 214 | 215
Participants | 9 | 10

ADVERSE EVENTS:
Time Frame: Serious and Other (Not Including Serious)Adverse Events (AEs) were collected from first dose of study drug up to 28days after last dose of study drug taken (up to data cut-off (15 Jan 2021)), approximately 2 years.
Arm/Group | HS-10296 | Gefitinib
All-Cause Mortality (participants affected / at risk) | 54/214 | 69/215
Serious Adverse Events (participants affected / at risk) | 47/214 | 46/215
Other Adverse Events (participants affected / at risk) | 211/214 | 213/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HS-10296 (N=214) | Gefitinib (N=215)
Pneumonia (Infections and infestations) | 6 (6) | 8 (8)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Skin infections (Infections and infestations) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 9 (9)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 2 (2)
Liver function injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Spontaneous pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Increased alanine aminotransferase (Investigations) | 0 (0) | 4 (4)
Increased aspartate aminotransferase (Investigations) | 0 (0) | 4 (4)
Increased aminotransferases (Investigations) | 0 (0) | 1 (1)
Decreased white blood cell count (Investigations) | 1 (1) | 0 (0)
Decreased neutrophil count (Investigations) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Acute cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Coronary atherosclerosis (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Cardiorespiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Ureteral stones (Renal and urinary disorders) | 1 (1) | 1 (1)
Impairment of renal function (Renal and urinary disorders) | 0 (0) | 1 (1)
Difficulty urinating (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humeral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Complications of hepatobiliary surgery (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoproteinemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Completed suicide (Nervous system disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Venous thrombosis of extremities (Vascular disorders) | 3 (3) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Liver cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Rhegmatogenous retinal detachment (Eye disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HS-10296 (N=214) | Gefitinib (N=215)
Weight loss (Investigations) | 14 (14) | 35 (35)
Blood bilirubin increased (Investigations) | 18 (18) | 34 (34)
γ-glutamyl transferase increased (Investigations) | 19 (19) | 30 (30)
Blood creatine phosphokinase increased (Investigations) | 76 (76) | 20 (20)
QT interval prolonged (Investigations) | 23 (23) | 19 (19)
Platelet count decreased (Investigations) | 47 (47) | 17 (17)
Blood lactate dehydrogenase increased (Investigations) | 26 (26) | 14 (14)
Erythra (Skin and subcutaneous tissue disorders) | 50 (50) | 89 (89)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (14) | 26 (26)
Dental ulcer (Gastrointestinal disorders) | 22 (22) | 21 (21)
Nausea (Gastrointestinal disorders) | 23 (23) | 20 (20)
Emesis (Gastrointestinal disorders) | 26 (26) | 11 (11)
Upper respiratory infection (Infections and infestations) | 41 (41) | 26 (26)
Hypokalemia (Metabolism and nutrition disorders) | 19 (19) | 33 (33)
Hypoalbuminemia (Metabolism and nutrition disorders) | 15 (15) | 23 (23)
Anemia (Blood and lymphatic system disorders) | 43 (43) | 21 (21)
Bound bilirubin increased (Investigations) | 7 (7) | 21 (21)
Blood in urine (Investigations) | 14 (14) | 16 (16)
Serum creatinine increased i (Investigations) | 11 (11) | 14 (14)
White blood cells in urine (Investigations) | 9 (9) | 12 (12)
Weight gain (Investigations) | 17 (17) | 11 (11)
Blood urea increased (Investigations) | 16 (16) | 11 (11)
Serum alkaline phosphatase increased (Investigations) | 15 (15) | 10 (10)
Decreased lymphocyte count (Investigations) | 11 (11) | 5 (5)
Increased Serum creatine phosphokinase MB (Investigations) | 13 (13) | 3 (3)
Constipation (Gastrointestinal disorders) | 20 (20) | 15 (15)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 11 (11)
Abdominal pain (Gastrointestinal disorders) | 20 (20) | 3 (3)
Pneumonia (Gastrointestinal disorders) | 15 (15) | 12 (12)
Hypocalcemia (Metabolism and nutrition disorders) | 19 (19) | 12 (12)
hyperuricemia (Metabolism and nutrition disorders) | 19 (19) | 10 (10)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 13 (13) | 7 (7)
weak (General disorders) | 12 (12) | 17 (17)
Influenza like illness (General disorders) | 7 (7) | 11 (11)
Sinus bradycardia (Cardiac disorders) | 8 (8) | 12 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 13 (13)
Proteinuria (Renal and urinary disorders) | 18 (18) | 19 (19)
Hematuria (Renal and urinary disorders) | 11 (11) | 18 (18)
Physical pain (Musculoskeletal and connective tissue disorders) | 15 (15) | 6 (6)
High blood pressure (Vascular disorders) | 15 (15) | 12 (12)
Insomnia (Psychiatric disorders) | 12 (12) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/68/NCT03849768/Prot_001.pdf
  • Statistical Analysis Plan (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/68/NCT03849768/SAP_002.pdf